CLINICAL TRIAL: NCT00728559
Title: Evaluation of Local Anlagesia Into the Trocar Site During Operative Laparosocpy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Ilan Atlas, MD Gynecologic Oncology Director, Poria Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lapmar1.CTIL
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2008-08

CONDITIONS: Pain
Keywords: laparoscopy; preemptive; postoperative; pain; trocar; site
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): preemptive trocar site analgesia
  Interventions: Drug: bupivacain 0.5%
- 2 (Experimental): trocar site pre skin closure analgesia
  Interventions: Drug: bupivacain 0.5%
- 3 (No Intervention): control

INTERVENTIONS:
Drug: bupivacain 0.5% — trocar site injection
  Other Names: marcaine
  Arms: 1; 2

SUMMARY:
In the literature there is conflicting data on administration of local analgesia in addition to the general anesthesia to the trocar sites during laparoscopy, We believe that adding local analgesia to the general anesthesia during laparoscopy is beneficial . the current study will evaluate prospectivly the impact of local analgesia on postoperative pain and recovery in patients undergoing operative laparoscopy

DETAILED DESCRIPTION:
Methods: this is a blinded prospective randomized study. After approval of IRB and informed consent 120 patients undergoing for laparoscopy will be randomized after the induction of general anesthesia into three groups: Group A will receive preemptive analgesia using 3-5 cc of 0,5 % marcaine at the beginning of the procedure. Group 2 will receive a local analgesia using 3-5 cc marcaine at the end of the procedure. Group 3 will be operated under general anesthesia only. The post operative pain and patient recovery will be assessed by the nurses during the hospitalization using a VAS (Visual Analog Scale) the total analgetic drugs will be noted and after the patients discharge the patient status and satisfaction will be evaluated by phone up to 2 wks

ELIGIBILITY:
Inclusion Criteria:

* Female older then 18 y/o

Exclusion Criteria:

* Allergy to marcaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
postoperative pain measured by VAS | 2 years

SECONDARY OUTCOMES:
total analgesics required, patient recovery, patient satisfaction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Atlas, MD, Study Chair — Ministry of Health, Israel
Locations (1):
- Poria Gov Hospital, Tiberias, Lower Galilee, Israel